CLINICAL TRIAL: NCT01553227
Title: Effect of Auto-trilevel Ventilator on Patients With Obstructive Sleep Apnea Hypopnea Syndrome and Obesity
Brief Title: Treatment for Obstructive Sleep Apnea Hypopnea Syndrome and Obesity Hypoventilation Syndrome (OHS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhang Xilong, The First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXZZ11-0726
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome
Keywords: OSAHS: Obstructive Sleep Apnea hypopnea Syndrome; OHS: Obesity Hypoventilation Syndrome; Auto-trilevel ventilation; BiPAP ventilation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome | interventions — Ventilators, Mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ventilator (Experimental): The overall purpose of this study is to determine the effects of auto-Trilevel ventilation on patients with OSAHS and OHS by comparison with BiPAP ventilation. The following parameters are compared such as apnea hypopnea index, lowest SPO2, arousal index, sleep efficiency, PaCO2, daytime sleepiness and so on.
  Interventions: Device: ventilator

INTERVENTIONS:
Device: ventilator — Noninvasive ventilation including fixed BiPAP ventilation and auto-trilevel ventilation. Using the same IPAP, treatment include one night with BiPAP ventilation mode 1, one night with BiPAP ventilation mode 2 and one night with auto-trilevel ventilation mode. Each treatment last 8 hours for each night.
  Other Names: Auto-trilevel ventilation

SUMMARY:
Sleep Apnea Hypopnea Syndrome (OSAHS), is common in patients with OHS, compared to single Obesity Hypoventilation Syndrome (OHS) or OSAHS ,patients with both of them are more susceptible to have serious hypoxia and carbon dioxide retention during sleep, and much more likely to result in pulmonary hypertension and cor-pulmonale.

At present, the most widely and valid method for these patients is the Bilevel Positive Airway Pressure (BiPAP) ventilation, while, recently, the investigators discovered a completely novel device, namely auto-trilevel Ventilator. In contrast to the traditional therapy, auto-trilevel Ventilator has a more flexible expiratory positive airway pressure (EPAP), with which it can removing residual obstructive sleep apnea hypopnea events and correcting hypercapnia without contradiction. Treated with auto-trilevel ventilator may delay the progression of disease and improve life quality. The overall purpose of this study is to determine the curative effects of auto-trilevel ventilators on patients with OHS and OSAHS.

DETAILED DESCRIPTION:
The main contradiction in treatment for OSAHS complicated OHS is how to improve hypercapnia because of narrower difference between inspiratory positive airway pressure (IPAP) and expiratory positive airway pressure (EPAP), and meanwhile to eliminate apnea and popnea events which may easily occur at the end of expiration For ordinary Bipap ventilator. If the IPAP is set to higher, the patients may feel discomfort, if the pressure difference between IPAP and EPAP is too narrow or the expiratory positive airway pressure (EPAP) too high, hypercapnia may occur. If the EPAP is too low, redusual apnea and hypopnea event may become common.

Auto-trilevel ventilation, with a lower airway pressure at the beginning of expiration to prevent hypercapnia and a higher airway pressure at the end of expiration to prevent residual apnea events, should be able to provide a novel ventilation mode with a higher efficacy and lower average airway pressure for OSAHS patients complicated with OHS. To prove the hypothesis, comparison is made between ordinary BiPAP and auto-Trilevel ventilation modes during treatment for patients with OSAHS and OHS.

In this study, the investigators compare the changes of related indexes (including apnea hypopnea index、minimal pulse oxygen saturation、arousal index, sleep quality,PaCO2 and sleepiness scores) before and after treatment. Meanwhile, curative effects will be compared between BiPAP and auto-Trilevel ventilation modes. The investigators will analyze the changes and then confirm our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative of the patient is willing and able to sign an approved informed consent and privacy protection authorization in the United States.
2. Subject is >18 years old.
3. Diagnosed OHS and OSAHS:
4. Expected to tolerate the ventilator therapy.

Exclusion Criteria:

1. Patient is currently enrolled in another clinical study which may confound the result of this study.
2. Patient for whom inform consent cannot be obtained.
3. Patients with a history of cerebrovascular accident within the 6 months prior to this study.
4. Patients with acute or chronic renal failure, diabetes and severe lung diseases.
5. Patients with unstable angina.
6. Patient who is of pregnant or during lactation period.
7. Patients with a history of injury or surgery within 6 months prior to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Effect of auto-trilevel ventilation on patients with OSAHS and OHS | Participants will be observed for the duration of hospital stay an expected average of 1 week
  The overall purpose of this study is to determine the effects of auto-trilevel ventilator on patients with OSAHS and OHS. The following parameters are compared such as apnea hypopnea index, lowest SPO2, arousal index, sleep efficiency, PaCO2, daytime sleepiness and so on.

CONTACTS AND LOCATIONS:
Overall Officials: xilong zhang, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China